CLINICAL TRIAL: NCT02044081
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Microbiology of C16G2 Administered in Multiple Oral Gel and/or Mouth Rinse Doses to Healthy Adult Subjects
Brief Title: Phase 2, Safety & Microbiology Study of C16G2 in Multiple Oral Gel &/or Mouth Rinse Doses to Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C3J13-201-01
Record Dates: First submitted 2014-01-09; First posted 2014-01-23 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mouth Rinse Administration (Other): Day 0, three consecutive C16G2 or placebo rinse administrations followed by three single C16G2 or placebo rinse administrations. Days 1 to 6 two additional C16G2 or placebo rinse administrations.
  Interventions: Drug: C16G2 Rinse; Drug: Placebo
- Dental Tray Gel Administration (Other): Day 0, two C16G2 or placebo gel dental tray applications and four C16G2 or placebo rinse administrations. Days 1 to 6, two C16G2 or placebo dental tray applications and two C16G2 or placebo rinse administrations.
  Interventions: Drug: C16G2 Rinse; Drug: Placebo; Drug: C16G2 Gel
- Electric Toothbrush Gel Application (Other): Day 0, four C16G2 or placebo gel administrations applied with an electric toothbrush and four C16G2 or placebo rinse administrations. Days 1 to 6, two C16G2 or placebo gel administrations applied with a electric toothbrush and two C16G2 or placebo rinse administrations.
  Interventions: Drug: C16G2 Rinse; Drug: Placebo; Drug: C16G2 Gel
- Manual Toothbrush Gel Application (Other): Day 0, four C16G2 or Placebo gel administrations applied with a manual toothbrush and four C16G2 or Placebo rinse administrations. Days 1 to 6, two C16G2 or Placebo gel administrations applied with a electric toothbrush and two C16G2 or Placebo rinse administrations.
  Interventions: Drug: C16G2 Rinse; Drug: Placebo; Drug: C16G2 Gel

INTERVENTIONS:
Drug: C16G2 Rinse — Active rinses are 1.6 mg/mL C16G2.
Drug: Placebo — Placebo is the vehicle without C16G2
Drug: C16G2 Gel — Active C16G2 Gel is 3.2 mg/mL
  Arms: Dental Tray Gel Administration; Electric Toothbrush Gel Application; Manual Toothbrush Gel Application

SUMMARY:
The focus of the study is to evaluate the safety of multiple study drug administrations and the study drug selectively reducing or eliminating a specific bacteria in the mouth. It will compare a liquid and gel product applied in different modes.

DETAILED DESCRIPTION:
The study will evaluate the safety of multiple study drug administrations as assessed by adverse event monitoring, oral cavity assessments, targeted physical exams and vital signs. The study will also assess the study drug's ability to selectively reduce or eliminate specific bacteria in the mouth by comparing a liquid and gel product applied in different modes, such as mouth rinse administration and gel application using a dental tray, electric toothbrush or manual toothbrush administered over 7 consecutive days. Subjects will be followed for approximately 8 days after the last study drug administration for safety and microbiology.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to participate if they meet the following criteria:

* Males and females, 18-75 years of age, inclusive, at the time the Informed Consent Form is signed
* Female subjects of childbearing potential, defined as not surgically sterile or at least two (2) years postmenopausal, must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, monogamous relationship with same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit.
* Male subjects only: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination.
* Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (extraoral, head and neck) during Screening
* Have a minimum of six unrestored bicuspids and molars with less than 50% of molars and bicuspids having restorations, crowns, sealants or are missing
* Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
* Demonstrated ability to swish 10 mL of water for 4 minutes
* Have a salivary and dental plaque S. mutans of 2.0 x 10^4 colony forming unit (CFU)s/mL or greater at Screening using mitis salivarius-bacitracin (MSB) agar plating
* Willing to refrain from using non-study dentifrice and other non-study oral care products during the study
* Willing to postpone elective dental procedures (e.g. dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
* Able to understand and sign the Informed Consent Form prior to initiation of study procedures
* Able to communicate with the Investigator/study site personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

Subjects are excluded from participation if any of the following apply:

* Advanced periodontal disease
* Active caries lesion(s) within 30 days prior to study drug administration (confirmed by dental examination and standard radiographs).
* Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
* Pathologic lesions of the oral cavity (suspicious or confirmed)
* Full or partial dentures, or orthodontic appliances, e.g. night guards, permanent retainers
* Impaired salivary function (unable to provide 2 mL of stimulated saliva within 5 minutes)
* Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, within 30 days prior to Screening
* Medical history indicating the woman is pregnant, breastfeeding/lactating or she has a positive urine pregnancy test
* Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
* Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of multiple C16G2 Gel and/or C16G2 Rinse administrations in healthy adult subjects. | Screening, Baseline, Days 1-7, & Day 14
  Safety will be assessed by comparing the incidence and duration of adverse events, clinically significant changes in vital signs, oral cavity assessments and targeted physical exams (C16G2 subjects in the four study arms vs. placebo).

SECONDARY OUTCOMES:
To assess the targeted antimicrobial activity of C16G2 gel and rinse applications as measured by a reduction of dental plaque and salivary Streptococcus mutans (S. mutans). | Screening, Baseline, Days 1, 7 & 14
  Saliva and dental plaque samples will be assessed at screening and Days 1, 7 and 14 for S. mutans (C16G2 subjects in the four study arms vs. placebo).
To assess total bacteria in dental plaque and saliva post-study drug. administration | Screening, Baseline, Days 1, 7 & 14
  Total bacteria will be assessed at screening, baseline and Days 1, 7 and 14 (C16G2 subjects in the four study arms vs. placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Marberger, DDS, Principal Investigator — Jean Brown Research
Locations (2):
- United States (2):
  - Plaza West II Dental Group, Kalispell, Montana
  - Jean Brown Research, Salt Lake City, Utah